CLINICAL TRIAL: NCT07281625
Title: A Randomized Controlled Trial Comparing Surgical Outcomes of Decompressive Laminectomy Versus Decompressive Laminectomy With Transpedicular Screw Fixation in Multilevel Lumbar Spinal Stenosis
Brief Title: Decompressive Laminectomy Versus Laminectomy With Transpedicular Fixation in Lumbar Spinal Stenosis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Punjab Health Care Commission (Other)
Responsible Party: Principal Investigator, Hira Umar, Doctor, Services Institute of Medical Sciences, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHL-LSS-Trial
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-10

CONDITIONS: Lumbar Spinal Stenosis
Keywords: laminectomy; spinal stenosis; lumbar fusion; VAS pain score
MeSH Terms: conditions — Spinal Stenosis | interventions — Laminectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decompressive Laminectomy Only (Active Comparator): Surgical decompressive laminectomy performed without instrumented fixation in patients with multilevel lumbar spinal stenosis.
  Interventions: Procedure: Decompressive Laminectomy; Procedure: Decompressive Laminectomy With Transpedicular Screw Fixation
- Laminectomy With Transpedicular Screw Fixation (Experimental): Surgical decompressive laminectomy combined with transpedicular screw fixation to provide additional spinal stability in patients with multilevel lumbar spinal stenosis.
  Interventions: Procedure: Decompressive Laminectomy; Procedure: Decompressive Laminectomy With Transpedicular Screw Fixation

INTERVENTIONS:
Procedure: Decompressive Laminectomy — Surgical removal of the vertebral lamina to decompress the spinal canal in patients with multilevel lumbar spinal stenosis. No instrumentation or fixation is applied.
Procedure: Decompressive Laminectomy With Transpedicular Screw Fixation — Surgical decompression via laminectomy combined with spinal stabilization using transpedicular pedicle screws for multilevel lumbar spinal stenosis to prevent postoperative instability and provide bony fusion.

SUMMARY:
Lumbar spinal stenosis is a condition where the spinal canal becomes narrowed and can cause symptoms such as back pain, numbness, leg pain, and difficulty walking. Surgery is often considered when symptoms do not improve with medical treatment.

This study will compare two types of surgery used to treat lumbar spinal stenosis: decompressive laminectomy alone and decompressive laminectomy with transpedicular screw fixation. Patients will be randomly assigned to one of the two surgical options.

The purpose of this study is to determine which approach provides better pain relief, improved function, fewer complications, and better spinal stability after surgery.

DETAILED DESCRIPTION:
Lumbar spinal stenosis (LSS) is a common degenerative spinal disorder causing neurogenic claudication, back pain, radiculopathy, and functional limitation. Multilevel stenosis is frequently associated with degenerative disc disease and facet joint hypertrophy. Decompressive laminectomy is a widely performed procedure; however, concerns exist regarding postoperative instability, which may affect long-term outcomes. Instrumented fixation using transpedicular screws may provide stability but also increases operative time, surgical risk, and healthcare cost.

This randomized controlled trial will be conducted at the Department of Neurosurgery, Services Hospital Lahore, over a six-month period. A total of 60 participants aged 30-60 years with MRI-confirmed multilevel lumbar spinal stenosis who have failed six weeks of conservative treatment will be enrolled using consecutive sampling and randomized into two equal study groups. Group A will undergo decompressive laminectomy alone, while Group B will undergo decompressive laminectomy with transpedicular screw fixation.

b2bf342f-1787-4c2e-828b-e000ffb…

Outcome measures will include operative time, postoperative complications, length of hospital stay, pain assessed using the Visual Analog Scale (VAS) at baseline, day 7, and 3 months, and functional status assessed using the Oswestry Disability Index (ODI) at baseline and 3 months. Postoperative radiographs will be used to evaluate spinal stability and bony fusion at 3 months.

b2bf342f-1787-4c2e-828b-e000ffb…

Data will be analyzed using SPSS version 25. Continuous variables will be presented as mean ± standard deviation and analyzed using an independent sample t-test. Categorical variables will be compared using the chi-square test, with a significance threshold of p ≤ 0.05. The study aims to evaluate whether decompression alone or decompression with transpedicular fixation results in superior clinical and radiological outcomes.

b2bf342f-1787-4c2e-828b-e000ffb…

ELIGIBILITY:
Inclusion Criteria:

* Age 30-60 years
* Diagnosis of lumbar spinal stenosis based on MRI criteria (anteroposterior canal diameter <10-15 mm or cross-sectional area <75-145 mm²)
* Multilevel disc herniation
* Degenerative disc disease with Pfirrmann grade 3-5 on T2-weighted MRI
* Failure of at least six weeks of conservative treatment

Exclusion Criteria:

* Previous history of lumbar spine surgery
* Spinal malignancy
* Congenital lumbar spinal stenosis, scoliosis, or kyphoscoliosis
* Lumbar spondylolisthesis grade 3-5
* Significant comorbidities including diabetes mellitus or ischemic heart disease

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Oswestry Disability Index (ODI) | Baseline and 3 months after surgery
  Functional disability will be assessed using the Oswestry Disability Index (ODI), recorded preoperatively and at 3-month follow-up to measure improvement in functional outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hira Umar, MBBS, Principal Investigator — SIMS
Locations (1):
- Services Institute of Medical Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Plans for sharing individual participant data have not yet been finalized. Data sharing may be limited by institutional policy, ethical requirements, and patient confidentiality considerations. If a data-sharing framework is approved in the future, the plan will be updated in this record.